CLINICAL TRIAL: NCT02132325
Title: Phase I/IIA: Dignity Therapy/Life Plan in Patients With Pancreatic or Advanced Lung Cancer
Brief Title: Dignity Therapy/Life Plan in Patients With Pancreatic or Advanced Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ann (Ann Marie) M. Dose, R.N., Ph.D., Clinical Nurse Researcher, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-001857
Record Dates: First submitted 2014-05-01; First posted 2014-05-07 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Pancreatic Cancer; Non-Small-Cell Lung Cancer
Keywords: Pancreatic Cancer; Dignity Therapy; Palliative Care; Advanced Lung Cancer; Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Dignity Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dignity Therapy (Experimental)
  Interventions: Behavioral: Dignity Therapy

INTERVENTIONS:
Behavioral: Dignity Therapy — Dignity Therapy/Life Plan will be provided by an advanced practice nurse or chaplain (APN/Chap), who has undergone training in provision of Dignity Therapy (offered through a 3-day group workshop by Dr. Harvey Chochinov).

SUMMARY:
This study will evaluate feasibility and acceptability of providing the Dignity Therapy/Life Plan intervention to pancreatic or advanced lung cancer patients presenting for treatment in the outpatient medical oncology setting. Investigators hypothesize that providing dignity therapy to this population will be feasible.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Undergoing chemotherapy for pancreatic adenocarcinoma or advanced NSCLC (pancreatic arm closed)
* English-speaking
* Cognitively intact, per clinician judgment, as documented in electronic medical record (EMR)

Exclusion Criteria:

* Currently receiving hospice or palliative care services
* Concurrent diagnosis of delirium or dementia, per medical record
* Diagnosis of major depression disorder, acute anxiety disorder or schizophrenia per medical record
* Participating in other psychosocial intervention research studies.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-04; Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Change in level of distress as measured by distress scores on the Distress Thermometer | Baseline & at the end of the dignity therapy intervention (approximately 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Marie Dose, PhD, RN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
A clean, deidentified data set will be made available to qualified requestors at study completion/dissemination.